CLINICAL TRIAL: NCT02274987
Title: A Pilot Trial Testing the Clinical Benefit of Using Molecular Profiling to Determine an Individualized Treatment Plan in Children With Newly Diagnosed DIPG
Brief Title: Molecular Profiling for Individualized Treatment Plan for DIPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Associate Adjunct Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNOC 003; 14082 (Other: University of California, San Francisco)
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Diffuse Intrinsic Pontine Glioma (DIPG)
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The treatment plan for each patient is individualized and different depending on what the Specialized Tumor Board recommends depending on the molecular profile of the patient's tumor.
  Interventions: Other: Specialized tumor board recommendation; Radiation: Standard radiation therapy

INTERVENTIONS:
Other: Specialized tumor board recommendation — A combination of up to four FDA approved drugs based on the molecular profile of the patient's tumor as determined by gene expression analysis, WES and predictive modeling.
Radiation: Standard radiation therapy — Initial therapy will consist of standard radiation therapy per institutional guidelines followed by molecular based therapy with FDA approved drugs.

SUMMARY:
This is a single arm multi-center pilot trial within the Pacific Pediatric Neuro-Oncology Consortium (PNOC). The current study will use a new treatment approach based on each patient's tumor genomic profiling consisting of whole exome sequencing and RNA sequencing as well as predictive modeling.

DETAILED DESCRIPTION:
The current study will test whether patients gain a clinical benefit from such a treatment approach by comparing overall survival at 12 months (OS12) to historical controls. Newly diagnosed patients will receive an individualized treatment recommendation including up to four FDA approved drugs based on the molecular profile of the patient's tumor as determined by gene expression analysis, Whole-exome sequencing (WES) and predictive modeling, age of the patient and other existing medical conditions. Initial therapy will consist of standard radiation therapy per institutional guidelines followed by molecular based therapy with FDA approved drugs.

ELIGIBILITY:
Inclusion Criteria for Newly Diagnosed Patients with diffuse intrinsic pontine glioma (DIPG):

* Diagnosis: Patients with newly diagnosed DIPG, defined as tumors with a pontine epicenter and diffuse involvement of the pons who undergo a biopsy are eligible. Patients with disseminated disease are not eligible, and MRI of the spine must be performed if disseminated disease is suspected by the treating physician.
* Enrollment within 28 days of the date of radiographic diagnosis.
* Age ≤ 25 years
* Karnofsky score ≥ 50 for patients ≥ 16 years of age and Lansky score ≥ 50 for patients ≤15 years of age. Patients who are unable to walk because of paralysis but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score .
* Organ Function Requirements:
* Adequate Bone Marrow Function Defined as:
* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm 3
* Platelet count ≥ 100,000/mm 3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin ≥ 8 g/dl (can be transfusion dependent)
* Adequate Renal Function Defined as:

Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70ml/min/1.73 m 2 OR a serum creatinine within normal limits based on age/gender as follows:

Maximum Serum Creatinine (mg/dL)

Age Male Female 3 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4

The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the United States Centers for Disease Control and Prevention (CDC).

* Organ Function Requirements cont.
* Adequate Liver Function Defined as:
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvic transaminase (SGPT) (ALT) ≤ 110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
* Serum albumin ≥ 2 g/dL
* The effects of the current treatment paradigm on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception: hormonal or barrier method of birth control; abstinence prior to study entry and for the duration of study participation, and 30 days after completion of study drug administration. Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 30 days after completion of study drug administration
* Adequate Neurologic Function Defined as:
* Patients with seizure disorder may be enrolled if seizures are well controlled.
* Ability by patient or parent/legal guardian (for patients under 18 years of age) to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria for Newly Diagnosed Patients with DIPG:

* Patients who are currently taking any anti-cancer directed therapy. Steroids are not considered anti-cancer therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy.
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
To determine OS12 of children with newly diagnosed DIPG that are being treated based on a specialized tumor board recommendation which is based on RNA based expression analysis, WES and predictive modeling. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol